CLINICAL TRIAL: NCT02232373
Title: A Pilot Double Blind, Randomised, Placebo Controlled Trial of the Effect of a Diet Low in Poorly Digested Carbohydrates on Symptoms of Post-infective Bowel Dysfunction
Brief Title: Campylobacter Enteritis and PI-BD: Dietary Reduction in Carbohydrates
Acronym: CEDRIC
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Failure to recruit
Sponsor: University of Nottingham (Other)
Collaborators: Nottingham University Hospitals NHS Trust (Other); King's College London (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: UoN14048; 14GA012 (Other: Nottingham University Hospitals NHS Trust)
Record Dates: First submitted 2014-09-02; First posted 2014-09-05 (Estimated); Last update posted 2016-05-13 (Estimated); Status verified 2016-05

CONDITIONS: Post-infective Bowel Dysfunction; Functional Gastrointestinal Disorders
Keywords: FODMAPs; microbiota; oligofructose; IBS; Irritable bowel syndrome
MeSH Terms: conditions — Gastrointestinal Diseases; Irritable Bowel Syndrome | interventions — maltodextrin; oligofructose

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Normal FODMAP arm (Sham Comparator): Low FODMAP dietary advice; participants to supplement diet with oligofructose, a poorly digested carbohydrate that will restore FODMAP content to the diet.
  Interventions: Behavioral: low FODMAP dietary advice; Dietary Supplement: Oligofructose
- Low FODMAP arm (Experimental): Low FODMAP dietary advice; participants to supplement with maltodextrin (easily digestible carbohydrate)
  Interventions: Behavioral: low FODMAP dietary advice; Dietary Supplement: Maltodextrin

INTERVENTIONS:
Behavioral: low FODMAP dietary advice — An education session with a specialist dietitian, and provision of written advice, on how to follow the low FODMAP diet. Second session after one month on re-introduction of FODMAP containing foods.
Dietary Supplement: Maltodextrin — Dietary supplementation with maltodextrin 5 grams twice daily for a month
  Arms: Low FODMAP arm
Dietary Supplement: Oligofructose — Dietary supplementation with oligofructose 5 grams twice daily for a month
  Other Names: OraftiP95
  Arms: Normal FODMAP arm

SUMMARY:
The purpose of the study is explore the issues that relate to testing a particular dietary treatment, the low FODMAP diet, in a randomised trial using an appropriate control diet with which to compare it. In this trial the investigators will look at its effect on symptoms of people with persistent disturbance in their bowel pattern 3 months after an intestinal infection with Campylobacter.

The investigators will also look at the changes in gut bacteria that occur with the diet.

ELIGIBILITY:
Inclusion Criteria:

* Participation in the CERAMIC study (see linked protocol)
* On-going post infective bowel dysfunction (PI-BD) 3 months after confirmation of Campylobacter spp. in stool sample. This is defined as responding 'No' to the question "have your bowels returned to normal since your Campylobacter infection?"
* Will consent to use of data and samples acquired for CERAMIC in the analysis of CEDRIC

Exclusion Criteria:

As for CERAMIC study (so already confirmed)

* Pregnancy declared by the candidate
* History declared by the candidate of pre-existing gastrointestinal disorder, including but not limited to: Inflammatory Bowel Disease; Coeliac Disease; Pancreatitis; Gallstone disease (biliary colic, cholecystitis); Diverticulitis; Cancer of the gastrointestinal tract; Irritable Bowel Syndrome
* Reported history of previous resection of any part of the gastrointestinal tract other than appendix or gallbladder
* Intestinal stoma
* Habitual use of opiate analgesics likely to alter bowel function e.g. morphine
* Use of antibiotics in the preceding four weeks other than for treatment of index infection. Any condition where the candidate is likely to require a course of antibiotics in the next 3 months e.g. severe chronic respiratory disease, recurrent urinary tract infection, lower limb ulceration
* Inability to complete the symptom questionnaires e.g. cognitive dysfunction, limiting memory and understanding
* Anyone who in the opinion of the investigator is unlikely to be able to comply with the protocol e.g. cognitive dysfunction, chaotic lifestyle related to substance abuse

Addition criteria for CEDRIC study:

* Use of antibiotics or prescribed probiotics during the CERAMIC study
* Failure to provide research stool samples during CERAMIC study
* Dietary practice not compatible with safe implementation of the trial diet e.g.veganism
* Medical reasons for pre-existing controlled diet that cannot be safely randomised e.g. end-stage kidney disease, diabetes

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2014-08; Primary Completion 2015-08 (Actual); Study Completion 2015-08 (Actual)

PRIMARY OUTCOMES:
Moderate or substantial improvement in irritable bowel syndrome (IBS) symptoms on IBS-GIS | 1 month after start of diet
  The IBS-GIS (Irritable Bowel Syndrome Global Improvement Score) is a validated 7-point balance scale to assess change in perception of symptoms in functional bowel disorders. Points 6 and 7 on the scale refer to moderate or substantial improvement. The outcome measure will be the proportion of participants in each group marking point 6 or 7 on the balance scale at this time point.

SECONDARY OUTCOMES:
Moderate or substantial improvement in IBS symptoms | 6 months after star of diet
  The IBS-GIS (Irritable Bowel Syndrome Global Improvement Score) is a validated 7-point balance scale to assess change in perception of symptoms in functional bowel disorders. Points 6 and 7 on the scale refer to moderate or substantial improvement. The outcome measure will be the proportion of participants in each group marking point 6 or 7 on the balance scale at this time point.
Adequate control of IBS symptoms | 1 month after start of diet
  Response to a yes/no question "Have your symptoms been adequately controlled?"
Adequate control of IBS symptoms | 6 months after start of diet
  Response to a yes/no question "Have your symptoms been adequately controlled?"
Percentage of days with loose stool | during last 14 days of dietary intervention
  Percentage of days with at least one stool of consistency type 6 or 7 on the Bristol stool form scale
Change from baseline in IBSS | 1 month after start of diet
  The IBSS (Irritable Bowel Symptom Severity Scale) is a validated composite score of symptoms in functional intestinal disorders
Change from baseline in IBSS | 6 months after start of diet
Change from baseline in fasting colonic volume | 1 month after start of diet
  This is a mechanistic endpoint. Colonic volume will be assessed by Magnetic Resonance Imaging at baseline and after intervention.
Change in fasting colonic gas volume | 1 month after start of diet
  This is a mechanistic endpoint. Colonic gas volume will be assessed by Magnetic Resonance Imaging at baseline and after intervention.
Change from baseline in stool concentration of Bifidobacteria | 1 month after start of diet
  This is a mechanistic endpoint, to assess changes in the microbiota caused by dietary intervention
Change from baseline in stool concentration of Bifidobacteria | 6 months after start of diet
  This is a mechanistic endpoint, to assess changes in the microbiota caused by dietary intervention

OTHER OUTCOMES:
Change from baseline in EQ-5D-5L score | 1 month after start of diet
  The EQ5D is a validated questionnaire to measure quality of life
Change from baseline in EQ-5D-5L score | 6 months after start of diet
Change from baseline in stool concentration of short-chain fatty acids | 1 month after start of diet
Change from baseline in stool concentration of short-chain fatty acids | 6 months after start of diet
Change from baseline in other clades of stool microbiota | 1 month after start of diet
  This will be exploratory work to assess the effect of the diet on other constituents of the stool microbiota
Change from baseline in other clades of stool microbiota | 6 months after start of diet

CONTACTS AND LOCATIONS:
Overall Officials: Giles AD Major, BM BCh MRCP, Principal Investigator — University of Nottingham; Robin C Spiller, PhD FRCP, Study Chair — University of Nottingham
Locations (1):
- University of Nottingham, Nottingham, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Departmental website — http://www.nddcbru.org.uk